CLINICAL TRIAL: NCT02045082
Title: Comparison Between the Sensibility of the Flocked Swab and the Traditional Fiber Swab for the Diagnosis of the Herpes Simplex Epithelial Keratitis
Brief Title: The Flocked Swab and the Traditional Fiber Swab for the Diagnosis of the Herpes Simplex Epithelial Keratitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: DR-002-1399, 2012-1649
Record Dates: First submitted 2014-01-21; First posted 2014-01-24 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Herpes Simplex Keratitis
Keywords: Flocked swab; Traditional fiber swab; Herpes simplex epithelial keratitis; Quantitative PCR
MeSH Terms: conditions — Keratitis, Herpetic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flocked swab (Copan 519CS01) (Experimental): Sampling of the cornea by the flocked swab
  Interventions: Procedure: Corneal sampling
- Traditionnal fiber swab (Copan 164KS01) (Experimental): Sampling of the cornea by the traditional finer swab
  Interventions: Procedure: Corneal sampling

INTERVENTIONS:
Procedure: Corneal sampling — Slit lamp corneal sampling with a Swab

SUMMARY:
The purpose of this study is to compare a corneal sampling realized by a flocked swab (flocked swab regular 519CS01) with a sampling by traditional fiber swab (Copan regular swab 164KS01 in polyester). Their impact on the sensibility of the viral culture in the Herpes simplex epithelial keratitis will be the primary objective of this study.

DETAILED DESCRIPTION:
In our center, the flocked swabs became an important tool in the corneal sampling for viral keratitis, replacing rightly or wrongly the former traditional fibers swab. No research was specifically designed to study the corneal taking with these swabs. Nevertheless, numerous reasons would motivate it, because of the peculiarities in ophthalmology: the corneal sampling has to be made with the slit lamp rather than in a macroscopic manner; the corneal lesion are often millimetre-length and confined; the histology of the cornea is unique and compares only imperfectly with other structures of the human body like the nasal mucosa. In these circumstances, the properties of the stalk (rigidity, length) and of its extremity (roughness, textures, absorbance) can influence the quality of the sampling and the final result of the culture.

ELIGIBILITY:
Inclusion Criteria:

* Slit lamp signs at the initial examination that are compatible with an Herpes simplex epithelial keratitis (Herpes simplex dendrite, herpes simplex geographic ulcer)

Exclusion Criteria:

* Topical or systemic antiviral Therapy during the last 14 days Patient with Herpes simplex stromal keratitis without epithelial involvement Herpetic lesion outside the cornea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Result of the culture | 1 month after the initial visit
  The result can be Positive or negative for Herpes simplex virus (HSV). Even if the result will be available in less than 1 week by the clinician after the culture, the research team will collect the data 1 month in average after the initial visit.

SECONDARY OUTCOMES:
Time before positivity of the culture | 1 month after the initial visit
  If the culture is positive for Herpes simplex virus, what is the time lapse(in day) before the culture became positive. The research team will collect the data 1 month in average after the initial visit by examining the microbiologic data of the laboratory.
Viral load concentration | 1 month after the initial visit
  Quantitative polymerase chain reaction (PCR) will be on a part of the sampling 1 month after the initial visit. The result will be the concentration of virus in number/ml detected in the sampling

CONTACTS AND LOCATIONS:
Overall Officials: Patricia-Ann Laughrea, MD, CRMC(C), Principal Investigator — Centre de recherche du CHU de Québec; Université Laval
Locations (1):
- Centre universitaire d'ophtalmologie, Hôpital du Saint-Sacrement, CHU de Québec, Québec, Quebec, Canada